CLINICAL TRIAL: NCT06280443
Title: Epidemiological Study of Sarcopenia in Patients With Chronic Lung Diseases: A Prospective Registry Cohort Study
Brief Title: Sarcopenia in Chronic Lung Diseases
Status: Recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Pin-Kuei Fu, MD, PhD, Principal Investigator, Taichung Veterans General Hospital
Other Study IDs: CE22407B
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Sarcopenia; COPD; Asthma; ILD
MeSH Terms: conditions — Sarcopenia; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inclusion criteria A)Outpatients with COPD (chronic obstructive pulmonary disease) or ILD (interstitial lung disease) from department of Chest medicine in Taichung Veterans General Hospital, judged by the doctor that they do not need hospitalization or emergent treatment.

B) Patients who agree to provide the ID card number to the research team for usage as a link to the National Health Insurance research database and Health bank to explore the continuity of care and the use of medical resources

DETAILED DESCRIPTION:
This study is a prospective, multi-center, and non-invasive cohort study. All participants are diagnosed with Asthma, COPD and ILD. We use SARC-Calf questionnaire, Frailty questionnaire and Grip strength as a tool for prescreen. According to the 2019 Asian Sarcopenia Consensus, participants are examined by SARC-Calf questionnaire, grip strength test and a physical performance test, including sit-stand test, short physical performance battery (SPPB), gait speed test and six-minute walk test. Bioelectrical impedance analysis (BIA) and Dual-energy X-ray absorptiometry (DXA) are applied to all participants by to analyze body composition. Participants are further classified into no Sarcopenia group, Sarcopenia group, and severe Sarcopenia group to derive the prevalence.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with COPD (chronic obstructive pulmonary disease) or ILD (interstitial lung disease) from department of Chest medicine in Taichung Veterans General Hospital, judged by the doctor that they do not need hospitalization or emergent treatment.
2. Those who meet the conditions for frailty diagnosis after assessment by the Frailty Scale
3. Patients who agree to provide the ID card number to the research team for usage as a link to the National Health Insurance research database and Health bank to explore the continuity of care and the use of medical resources
4. Age>=20

Exclusion Criteria:

1. Patients who refuse to sign the consent form
2. Patients who are bed ridden or unable to walk due to physical disabilities
3. Patients with terminal cancer or human acquired immunodeficiency syndrome
4. Patients with edema (pitting edema +2)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Baseline demographic characteristic, health behavior and exercise habits are collected by questionnaires.The main disease diagnosis, medication, clinical assessment questionnaire or biochemical examination and radiological examination results in outpatient visit are collected.
  * According to the 2019 Asian Sarcopenia Consensus, participants are examined by SARC-Calf questionnaire, grip strength test, frailty index and a physical performance test,including sit-stand test, short physical performance battery (SPPB), gait speed test and six-minute walk test. Afterward, bioelectrical impedance analysis (BIA) are applied to all participants by to analyze body composition. Participants are classified into Sarcopenia group and severe Sarcopenia group.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-10-13 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
sarcopenia rate | 1 year
  The proportion of sarcopenia diagnosis in patients with chronic lung diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan